CLINICAL TRIAL: NCT02186145
Title: Single Blind Randomized Study of Efficacy and Safety of Vaginal Cream With Association of Metronidazole, Nystatin and Dexamethasone in the Treatment of Bacterial and Fungal Vaginal Infections
Brief Title: Efficacy and Safety Study of Metronidazole, Nystatin and Dexamethasone Combination Therapy in Bacterial and Fungal Vaginal Infections
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marjan Industria e Comercio ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MJ 3002-13
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2014-07

CONDITIONS: Bacterial Vaginosis; Fungal Vaginal Infections
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Nystatin; Dexamethasone; Metronidazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Association of metronidazole; nystatin and dexamethasone (Experimental): Intravaginal cream containing metronidazole (500 mg), nystatin ( 100.000 UI) and dexamethasone (0,32 mg) once a day. Period: 10 days.
  Interventions: Drug: Association of metronidazole; nystatin and dexamethasone
- Flagyl (Active Comparator): Vaginal cream of metronidazole 500 mg, nystatin 100.000 UI - once a day. Period: 10 days
  Interventions: Drug: Flagyl

INTERVENTIONS:
Drug: Association of metronidazole; nystatin and dexamethasone
  Arms: Association of metronidazole; nystatin and dexamethasone
Drug: Flagyl — Vaginal cream of metronidazole and nystatin
  Other Names: Flagyl-Nistatina (Sanofi Aventis)
  Arms: Flagyl

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of association of metronidazole, nystatin and dexamethasone in the treatment of bacterial and fungal vaginal infections.

ELIGIBILITY:
Inclusion Criteria:

* Post-menarche women and premenopausal women, between 18 and 50 years old;
* Diagnosis of bacterial vaginosis (Amsel criteria), fungal (positive KOH test)or mixed vaginal infection;
* Patients who have regular menstrual cycles (patients with regular menstrual cycles with intervals between 21 to 35 days, duration of 1 to 7 days)

Exclusion Criteria:

* Patients who have a known hypersensitivity to components of the formula ;
* Pregnant and lactating women ;
* Patients with other vaginal infections, such as infection by Trichomonas vaginalis , C. trachomatis, Neisseria gonorrhoeae , herpes or HPV.
* Knowledge of positive test result for human immunodeficiency virus ;
* Patients in treatment of cervical intraepithelial neoplasia or carcinoma of the cervix ;
* Patients who have undergone gynecological procedures in the month prior to inclusion (such as cauterization of the cervix , cervical biopsy, high-frequency surgery) ;
* Patients with other vaginal or vulvar conditions that may confound interpretation of clinical response;
* Patients who received intravaginal or systemic antimicrobial or antifungal therapy 14 days before randomization ;
* Patients on immunosuppressive medications (such as corticosteroids , cyclosporine , etc. ) ;
* Known or suspected cancer ;
* Participation in any experimental study or ingestion of any experimental drug 12 months before the start of this study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Therapeutic cure | Day 21-35
  Therapeutic cure which is based on a combination of clinical outcome and Gram's stain results (Nugentscore)/mycological eradication.

SECONDARY OUTCOMES:
Evaluation on vulvovaginal inflammation | 21 - 35 days
  Time resolution of symptoms; percentage of patients with Nugent score between 0-3; negative fungal culture; and subjective assessment of patients on the intensity of vulvar itching.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine of ABC (FMABC), Santo André, São Paulo, Brazil